CLINICAL TRIAL: NCT04737525
Title: The Influence of a Connective Tissue Graft Versus a Porcine-derived Membrane (Mucoderm) on the Aesthetic Outcome After Immediate Placement and Loading of a Tapered Dental Implant in the Anterior Maxilla. A Randomized Controlled Clinical Trial.
Brief Title: Connective Tissue Graft Versus a Porcine-derived Membrane (Mucoderm) After Immediate Placement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilniaus Implantologijos Centro (VIC) Klinika (Network)
Collaborators: Straumann Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS1418
Record Dates: First submitted 2021-01-15; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Immediate Implants
Keywords: Soft tissue grafting

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Immediate implant placement and temporization of tapered implants after tooth extraction with buccal augmentation using allogenic bone and porcine-derived membrane.
  Interventions: Device: Dental implant placement, bone and soft tissue augmentation on buccal site
- Control group (Experimental): Immediate implant placement and temporization of tapered implants after tooth extraction with buccal augmentation using allogenic bone and connective tissue grafting (CTG).
  Interventions: Device: Dental implant placement, bone and soft tissue augmentation on buccal site

INTERVENTIONS:
Device: Dental implant placement, bone and soft tissue augmentation on buccal site — 1. Atraumatic extraction
  2. Palatinal positioning of tapered implant (BLX) 3.75mm diameter
  3. 3-4 mm below vestibular gingival line or 1 mm below bone crest
  4. Implant placement
  5. Allogenic bone packing of the "jumping distance" and soft tissue grafting
  6. Connective tissue graft (CTG) or porcine-derived membrane
  7. Provisional restoration out of occlusion and mandibular movements
  8. X-ray

SUMMARY:
Esthetic outcome of immediate implant placement in fresh extraction sockets remains one of the biggest challenges in implant dentistry. Recently a method to preserve the peri-implant tissues was introduced using provisional restoration, allogenic bone and soft tissue thickening. However, the evidence that this immediate provisialisation with soft tissue grafting using different grafting materials results in constantly high Pink Esthetic scores, especially compared to the delayed loading approach is still lacking.

The aim of this clinical trial is to assess the esthetic outcome of immediate temporization of immediately placed and loaded tapered implants in fresh extraction sockets with bone and soft tissue augmentation, using either a connective tissue graft (CTG) or a porcine-derived membrane (Mucoderm) in maxillary anterior sites.

The secondary objectives are to investigate the influence of immediate loading on the success rate of tapered implants and crestal bone levels.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of at least 18 years of age
2. 1 implant per patient
3. Subject must have voluntarily signed the informed consent before any study related action, are willing and able to attend scheduled follow-up visits, and agree that the pseudonymized data will be collected and analyzed
4. Anterior single teeth (canines and incisors) in both jaws
5. Class I extraction socket (intact buccal wall) or Class II (1/3 of buccal wall)
6. No recession of gingival contour of tooth to be extracted
7. No periodontal bone loss of neighboring anterior teeth
8. No implants in neighboring teeth
9. Atraumatic extraction of the tooth with intact socket walls remaining

Exclusion Criteria:

1. Deep bite (severe II class)
2. Heavy smokers (more than 10 cigarettes/day)
3. Systemic disease (diabetes, osteoporosis)
4. Primary stability after implant placement not achieved
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2031-02-10 (Estimated)

PRIMARY OUTCOMES:
Aesthetic evaluation | Change from baseline, 1 year, 5 and 10 years after prosthetic delivery
  Pink esthetic score (PES) according to Fürhauser et al. 2005 Seven variables will be evaluated: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES is 14. For the PES assessment, frontal photographs will be taken using a digital camera with a flash strobe mounted on a tripod (Canon 350d, 3456×2304 pixel resolution). PES will be assessed at baseline (Final Prosthesis), 3- and 12-month visit.

SECONDARY OUTCOMES:
Recession of gingiva (REC) | Change from baseline, 1 year, 5 and 10 years after prosthetic delivery
  Position of the gingival/mucosal margin - recorded with a periodontal probe from the incisal edge to the margin at the zenith.

CONTACTS AND LOCATIONS:
Locations (1):
- VIC clinic, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No